CLINICAL TRIAL: NCT07161960
Title: Early Versus Delayed Cholecystectomy After Percutaneous Drainage in Moderate and Severe Cholecystitis (ESCAPE Trial)
Brief Title: Early Versus Delayed Cholecystectomy After Percutaneous Cholecystostomy in Moderate and Severe Cholecystitis (ESCAPE)
Acronym: ESCAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yada Suwan (Other)
Collaborators: Chiang Mai University (Other); Lampang Hospital (Other); Phrae Hospital (Unknown); Maharaj Nakorn Chiang Mai Hospital (Other)
Responsible Party: Sponsor-Investigator, Yada Suwan, Yada Suwan, Doctor of Medicine, Chiang Mai University
Organization: Chiang Mai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUR-2568-0197
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Acute Cholecystitis; Percutaneous Cholecystostomy; Laparoscopic Cholecystectomy
Keywords: Acute cholecystitis; Percutaneous cholecystostomy; Laparoscopic cholecystectomy; Early LC; Delay LC
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Laparoscopic Cholecystectomy (Experimental): The patients will undergo laparoscopic cholecystectomy (LC) within the same admission of PCC and after PCC for 72 hours, usually not more than 2 weeks.
  Interventions: Procedure: Laparoscopic cholecystectomy
- Delay Laparoscopic Cholecystectomy (Experimental): The patients will undergo laparoscopic cholecystectomy (LC) after 6 weeks from PCC insertion, avoiding active inflammation and swelling
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy is the definite treatment for acute cholecystitis. According to Tokyo Guideline 2018, the proper timing of delay LC remains unclear due to lack to proper evidence.

SUMMARY:
Abstract:

Acute cholecystitis (AC) is typically managed according to the 2018 Tokyo Guidelines, with treatment strategies determined by the severity of the disease, patient comorbidities, and hospital capabilities. In cases of moderate AC, treatment options include antibiotics with delayed laparoscopic cholecystectomy (LC), antibiotics with early LC, or antibiotics with percutaneous cholecystostomy (PCC) followed by delayed LC. However, the Toyo Guideline 2018 suggested that there is a lack of consensus regarding the optimal timing for surgery following PCC due to insufficient scientific evidence. In practice, delayed LC is often performed approximately 6 weeks after PCC insertion.

While PCC can serve as a treatment option before definite surgery, complications such as tube dislodgment, obstruction, and failure to ambulate are common, leading to further hospital admissions and increased comorbidities. The ESCAPE trial was conducted to evaluate the optimal timing for LC following PCC in moderate and severe forms of acute cholecystitis, with the goal of improving treatment standards and reducing complications associated with PCC retention. We hypothesize that early LC after PCC insertion will be a feasible and effective alternative.

Methods:

This prospective, randomized controlled trial enrolled patients diagnosed with moderate to severe acute cholecystitis who underwent PCC. Clinical manifestations and laboratory parameters were monitored for 72 hours following PCC insertion. Patients demonstrating clinical or laboratory improvement were subsequently randomized into two groups: early LC and delayed LC.

* Early LC group: Laparoscopic cholecystectomy was performed during the same hospitalization.
* Delayed LC group: Laparoscopic cholecystectomy was performed more than 6 weeks after PCC insertion.

The primary endpoint/outcome is comprehensive complication index (CCI) from PCC and LC. Secondary endpoints include Nasaar Difficulty Scoring, length of hospital stay, rate of subtotal cholecystectomy, rate of conversion to open cholecystectomy and incidence of bile duct injury.

Results and Discussion:

The results of this study will provide valuable insights into the timing of LC following PCC and may influence future treatment protocols for moderate and severe acute cholecystitis. By assessing the feasibility and safety of early LC after PCC insertion, the ESCAPE trial aims to reduce the burden of PCC-related complications and optimize patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The patients are diagnosed moderate or severe from of acute cholecystitis according to Tokyo Guideline 2018.
* PCC insertion was performed by body interventionists or surgeons.
* Laparoscopic cholecystectomy will be performed in Maharaj Nakorn Chiang Mai Hospital, Lampang Hospital and Phrae Hospital.
* Age equal or more than 20 years-old

Exclusion Criteria:

* The patients that suspected CBD stone and need to undergo EUS / ERCP.
* Coincidence perihepatic abscess or liver abscess
* The patients with active or severe underlying disease, whom specialists suggest to postpone an operation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index from PCC and LC | From enrollment to 3 months postoperative
  Comprehensive Complication Index (CCI)is a score derived from Clavien-Dindo Classification. In this study, the complications include both from Percutaneous Cholecystostomy (PCC) and from Laparoscopic Cholecystectomy (LC). The Clavien-Dindo Classification is ranging from 1 (any deviation from postoperative course) to 5 (death). CCI integrates all CD complications and weights its severity. CCI is ranging from 0 (no complication) to 100 (death).

SECONDARY OUTCOMES:
Nasaar Difficulty Scoring | During the operation
  Nasaar Difficulty Scoring is used to evaluate intraoperative finding of LC difficulty, determining by the surgeons who perform LC. The scores include 3 aspects; gallbladder, cystic pedicle and adhesion. In each aspect, the score is ranging from 1 (the easiest) to 4 (the hardest).
Length of Hospital Stay (LOS) | During enrollment to 3 months postoperative or date that complication resolves
  In the early LC group, LOS refers to the duration that the patients stays in the hospital for the treatment for acute cholecystitis. In the delay LC group, LOS refers to duration of the first admission (admit for PCC insertion), the admission for LC and other admissions that are associated with PCC retention or LC complication.
Rate of Conversion to Open Cholecystectomy | During the operation
Rate of Subtotal Cholecystectomy | During the operation
Incidence of Bile Duct Injury | During the operation to 3 months postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Chiang Mai University 110 Inthawarorot Road, Sri Phum, Mueang, Chiang Mai 50200, Thailand, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No
According to the ethic consideration by the committee of Research, Chiang Mai University, the identification and all treatment history will be reached by the researchers, data collectors and analyzers only to keep privacy for the participants.

REFERENCES:
- [Result] Yamazaki S, Shimizu A, Kubota K, Notake T, Yoshizawa T, Masuo H, Sakai H, Hosoda K, Hayashi H, Yasukawa K, Umemura K, Kamachi A, Goto T, Tomida H, Seki H, Shimura M, Soejima Y. Urgent versus elective laparoscopic cholecystectomy following percutaneous transhepatic gallbladder drainage for high-risk grade II acute cholecystitis. Asian J Surg. 2023 Jan;46(1):431-437. doi: 10.1016/j.asjsur.2022.05.046. Epub 2022 May 21. PMID 35610148
- [Result] Woodward SG, Rios-Diaz AJ, Zheng R, McPartland C, Tholey R, Tatarian T, Palazzo F. Finding the Most Favorable Timing for Cholecystectomy after Percutaneous Cholecystostomy Tube Placement: An Analysis of Institutional and National Data. J Am Coll Surg. 2021 Jan;232(1):55-64. doi: 10.1016/j.jamcollsurg.2020.10.010. Epub 2020 Oct 21. PMID 33098966
- [Result] Okamoto K, Suzuki K, Takada T, Strasberg SM, Asbun HJ, Endo I, Iwashita Y, Hibi T, Pitt HA, Umezawa A, Asai K, Han HS, Hwang TL, Mori Y, Yoon YS, Huang WS, Belli G, Dervenis C, Yokoe M, Kiriyama S, Itoi T, Jagannath P, Garden OJ, Miura F, Nakamura M, Horiguchi A, Wakabayashi G, Cherqui D, de Santibanes E, Shikata S, Noguchi Y, Ukai T, Higuchi R, Wada K, Honda G, Supe AN, Yoshida M, Mayumi T, Gouma DJ, Deziel DJ, Liau KH, Chen MF, Shibao K, Liu KH, Su CH, Chan ACW, Yoon DS, Choi IS, Jonas E, Chen XP, Fan ST, Ker CG, Gimenez ME, Kitano S, Inomata M, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018: flowchart for the management of acute cholecystitis. J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):55-72. doi: 10.1002/jhbp.516. Epub 2017 Dec 20. PMID 29045062
- [Result] Molavi I, Schellenberg A, Christian F. Clinical and operative outcomes of patients with acute cholecystitis who are treated initially with image-guided cholecystostomy. Can J Surg. 2018 Jun;61(3):195-199. doi: 10.1503/cjs.003517. PMID 29806817
- [Result] Bao J, Wang J, Shang H, Hao C, Liu J, Zhang D, Han S, Li Z. The choice of operation timing of laparoscopic cholecystectomy (LC) after percutaneous transhepatic gallbladder drainage (PTGBD) for acute cholecystitis: a retrospective clinical analysis. Ann Palliat Med. 2021 Aug;10(8):9096-9104. doi: 10.21037/apm-21-1906. PMID 34488395
- [Result] Lyu Y, Li T, Wang B, Cheng Y. Early laparoscopic cholecystectomy after percutaneous transhepatic gallbladder drainage for acute cholecystitis. Sci Rep. 2021 Jan 28;11(1):2516. doi: 10.1038/s41598-021-82089-4. PMID 33510242